CLINICAL TRIAL: NCT06022445
Title: Prospective Validation of CARPET Prognostic Model for Patients With Septic Shock After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Prospective Validation of CARPET Prognostic Model for Septic Shock After Allo-HSCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other); Second Hospital of Shanxi Medical University (Other); The Second Hospital of Hebei Medical University (Other); Shanghai Zhongshan Hospital (Other); Shanxi Dayi Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Guangzhou University of Chinese Medicine (Other); The First Affiliated Hospital of Zhengzhou University (Other); Peking Union Medical College (Other); First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking University Institute of Hematology, Peking University People's Hospital
Other Study IDs: PKUPH-model validation
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Stem Cell Transplant Complications
Keywords: septic shock; prognostic model; allogeneic hematopoietic stem cell transplant
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with septic shock after allo-HSCT: patients who underwent allo-HSCT and experienced septic shock
  Interventions: Other: CARPET prognostic model

INTERVENTIONS:
Other: CARPET prognostic model — For patients diagnosed with septic shock, we obtained the information in CARPET prognostic model including time of septic shock, albumin, bilirubin, PaO2/FiO2, lactate, and GFR. We calculated the CARPET risk score and the 28-day mortality probability according to CARPET logistic regression model.

SUMMARY:
Validation of CARPET prognostic model for septic shock after allo-HSCT: a multicenter, prospective, and cohort study

DETAILED DESCRIPTION:
A clinical prognostic model named CARPET model for septic shock after allo-HSCT has been developed and internally retrospectively validated. A multicenter, prospective cohort study is planned to validate this clinical prediction model again.

The equation of the prediction model for 28-day mortality was as follows:

Probability(28-day mortality)=(exp⁡(Y))/(1+exp⁡(Y)) where Y=2.343+1.328* Time of septic shock- 0.085* Albumin + 0.016 * Bilirubin-0.003*PaO2/FiO2 +0.127*Lactate- 0.011 * Glomerular filtration rate

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* underwent allo-HSCT
* diagnosed with septic shock

Exclusion Criteria:

* experienced septic shock before enrollment
* relapsed or progressed after HSCT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included patients diagnosed with septic shock after allo-HSCT. The clinical criteria of septic shock were sepsis as defined by suspected or documented infection and an acute increase of ≥ 2 SOFA points, together with vasopressor therapy (norepinephrine, dopamine, vasopressin, or any other vasopressor) needed to elevate mean arterial pressure ≥ 65 mmHg and lactate >2 mmol/L (18 mg/dL) despite adequate fluid resuscitation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  Dead or alive at day 28 after septic shock diagnosis

SECONDARY OUTCOMES:
ICU length of stay | up to 1 year
  Days in the ICU after septic shock diagnosis
90-day mortality | 90 days
  Dead or alive at day 90 after septic shock diagnosis
Time on ventilator | up to 1 year
  Days in need of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University Insititute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymised participant data will be made available to researchers upon reasonable request after termination and publication of the study.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the termination and publication of the study
Access Criteria: Reasonable request by researcher based on study protocol.